CLINICAL TRIAL: NCT03444428
Title: The Relationship Between Arterial Stiffness and Respiratory Failure: Using Motor Neurone Disease as a Paradigm to Assess the Consequence of Sleep Disordered Breathing on Arterial Stiffness
Brief Title: The Relationship Between Arterial Stiffness and Respiratory Failure in Motor Neurone Disease
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 210214 16/LO/1560
Record Dates: First submitted 2017-07-31; First posted 2018-02-23 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Motor Neurone Disease; Hypoxemia and/or Hypercapnia
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non Invasive Ventilation: * Age, height, weight
  * History and Physical Examination
  * Evaluation of dyspnoea: mMRC, Borg scale (Seated-Supine)
  * Amyotrophic lateral sclerosis functional rating scale (ALSFRS-R)
  * Sleep-Disordered Breathing in Neuromuscular Disease Questionnaire (SiNQ-5)
  * 24h Blood Pressure monitor
  * Spirometry - FEV1 and FVC
  * Respiratory muscle strength - MIP, MEP, and SNIP
  * Arterial Blood Gases
  * Carotid-femoral pulse wave velocity
  * Breath CO exhale
  Interventions: Other: Non Invasive Ventilation
- Without Non Invasive Ventilation: Age, height, weight
  * History and Physical Examination
  * Evaluation of dyspnoea: mMRC, Borg scale (Seated-Supine)
  * Amyotrophic lateral sclerosis functional rating scale (ALSFRS-R)
  * Sleep-Disordered Breathing in Neuromuscular Disease Questionnaire (SiNQ-5)
  * 24h Blood Pressure monitor
  * Spirometry - FEV1 and FVC
  * Respiratory muscle strength - MIP, MEP, and SNIP
  * Arterial Blood Gases
  * Carotid-femoral pulse wave velocity
  * Breath CO exhale
  Interventions: Other: Without Non Invasive Ventilation

INTERVENTIONS:
Other: Non Invasive Ventilation — Assessments for those participants who are being set up onto NIV
  Groups: Non Invasive Ventilation
Other: Without Non Invasive Ventilation — Assessments for those participants who are not being set up onto NIV
  Groups: Without Non Invasive Ventilation

SUMMARY:
* Patients with Motor Neurone Disease (MND) admitted to Lane Fox Unit /Royal Brompton Hospital and/or reviewed in Lane Fox Unit /Royal Brompton Hospital clinics and/or outreach review will be approached for participation in the study
* Physiological assessment and measurement of arterial stiffness will be performed in all patients at baseline and after the use of non invasive ventilation for 6 weeks.
* MND patients not requiring mechanical ventilation will serve as controls since non invasive ventilation cannot be withheld from MND patients in type II respiratory failure.
* Data will be analysed to look for differences between groups, relationships in baseline or change from baseline in respiratory physiological measures, inflammatory indices, breathlessness, and arterial stiffness.

  * Age, Height, Weight
  * History and Physical Examination
  * Evaluation of dysponea: mMRC, Borg Scale (Seated-Supine)
  * Amyotrophic lateral sclerosis functional rating scale (ALSFRS-R)
  * Sleep Disordered Breathing in Neuromuscular Disease Questionnaire (SiNQ-5)
  * 24 hour blood pressure monitor
  * Carotid-femoral pulse wave velocity
  * Respiratory Muscle Strength - Maximal Inspiratory Pressure, Maximal Expiratory Pressure, and Sniff Nasal Inspiratory Pressure
  * Spirometry - FEV1 and FVC
  * Arterial Blood Gas
  * CRP and fibrinogen (clinically)
  * Breathe CO exhale

DETAILED DESCRIPTION:
The stiffness of the arterial wall is highly relevant to cardiovascular disease. Large elastic arteries and smaller muscular conduit arteries become stiffer with ageing, a process that is accelerated in the presence of cardiovascular disease. Arterial stiffness increases also with various disease states, including hypertension, diabetes mellitus, obesity, smoking, hypercholesterolemia, and kidney disease. Numerous techniques have been developed to measure arterial stiffness, either in single vessels or in entire muscular arterial trees. These techniques have increasingly been shown to improve stratification of cardiovascular risk and risk reduction beyond that provided by conventional risk factors. Furthermore, large artery stiffness, measured via carotid-femoral pulse wave velocity, independently predicts the risk of cardiovascular events in both clinical and community-based cohorts.

Abnormalities in arterial stiffness have been noted in disorders characterized by hypoxia with or without hypercapnia. These abnormalities could be driven by the risk factors for those conditions (e.g. cigarette smoke, obesity). In COPD, all studies are consistent showing a significant increase in arterial stiffness compared with ex-smokers without airway obstruction and nonsmoker healthy control subjects. The severity of airway obstruction is consistently related to arterial stiffness in COPD. Furthermore, airflow limitation arising from cigarette smoking, but not airflow limitation in non-smokers, was associated with arterial stiffness in a general population independently of established risk factors. The presence of OSA was associated with higher arterial stiffness indices independent of major confounders. In this context, OSA is associated with increased arterial stiffness independent of blood pressure.

Non invasive ventilation has been shown to reduce arterial stiffness in obstructive sleep apnea. In particular, there are studies that have examined the impact of continuous positive airway pressure (CPAP) on arterial stiffness (measured with pulse wave velocity) in OSA patients. Other studies have examined changes in arterial stiffness (measured with other than pulse wave velocity method) after treatment of OSA with CPAP. Furthermore, to the best of our knowledge no investigation exists on the impact of non invasive bilevel positive airway pressure ventilation on arterial stiffness in neuromuscular disease.

The Lane Fox Unit, the UK's largest weaning, rehabilitation and home ventilation unit, is treating neuromuscular patients. In neuromuscular disease, especially in MND, confounding factors as obesity, cigarette smoke, hypertension, and diabetes mellitus can be excluded. This gives the opportunity to determine whether hypoxemia and/or hypercapnia alone cause arterial stiffness. Furthermore, in this pilot study it will be investigated whether non invasive ventilation has any effect on arterial stiffness in MND patients.

ELIGIBILITY:
Inclusion Criteria:

* MND diagnosis
* The ability to perform the respiratory function testing satisfactorily
* Stable clinical and functional state for at least four weeks before testing
* BMI 20-30 kg•m-2

Exclusion Criteria:

* Pregnancy
* Aged <18, >80
* Significant physical or psychiatric comorbidity that would prevent compliance with trial protocol
* Unstable clinical state
* Use of mechanical ventilation
* Cardiovascular disorders (history, physical examination)
* Known lung disease, such as asthma or COPD or any other cause of hypoxemia and/or hypercapnia but MND (history, physical examination, CXR review [High Resolution Computed Tomography if CXR is not compatible with neuromuscular disease alone])
* Airway obstruction (FEV1/FVC<0.75)
* Diabetes mellitus
* Obesity (BMI>30 kg•m-2)
* Smoking history (>10 pack∙years or active smoker)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Motor Neurone Disease
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Comparing the pulse wave velocity between MND patients with hypoxemia and/or hypercapnia to those MND Patients that do not have hypoxemia and/or hypercapnia | 6 weeks
  Is there a difference in pulse wave velocity between patients with MND who have and those who do not have hypoxemia and/or hypercapnia

SECONDARY OUTCOMES:
Comparison of pulse wave velocity values in MND patients to normal values | 6 weeks
  To clarify if there is an increased pulse wave velocity in MND patients and quantify whether patients are within predicted values or not against current evidenced literature
Comparison of pulse wave velocity pre-post non invasive ventilation in MND patients | 6 weeks
  Does NIV change pulse wave velocity in MND patients

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Murphy, Principal Investigator — Guys and St Thomas NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Guys and St Thomas NHS Trust, London
  - Royal Brompton and Harefield NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available